CLINICAL TRIAL: NCT03800316
Title: Synchronous Video (Telemedicine) Consulation in the Prehospital Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher S. Russi, Prinipal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-005054
Record Dates: First submitted 2018-12-10; First posted 2019-01-11 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: Emergencies; Prehospital; Telemedicine; Telehealth
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Synchronous Video Consultation (Experimental): Testing the feasibility of a synchronous video consultation in the field prior to emergency department arrival.
  Interventions: Device: Video Consultation

INTERVENTIONS:
Device: Video Consultation — Video consultation with emergency medicine physicians for patients that are critically ill prior to arrival in the ED

SUMMARY:
The study team aims to test connectivity metrics and follow patient outcomes using a new, innovative synchronous video technology in the prehospital setting in three distinct areas:

1. - 911 Calls
2. - Pediatric Critical Care Transport

Currently, paramedics and pediatric transport teams seek advice from physicians using a telephone. This project replaces the phone with video consultation where the physicians can directly interact with patients, paramedics and transport teams when care advice is needed.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Arrest
* Hemodynamically unstable trauma patients requiring resuscitation and airway management
* Trauma patients with altered mentation requiring airway management
* Acute stroke patients
* Medical patients that refuse transport for medical evaluation Pediatric Intensive Care Telemedicine Program
* Complex clinical situations where paramedic teams need immediate management guidance
* Critically ill pediatric patients requiring evaluation/stabilization for interfacility transport
* Pediatric patients requiring intervention for respiratory failure
* Pediatric patients with ongoing seizures and/or neurological abnormalities
* Hemodynamically unstable patients
* Complex clinical situations requiring medical control guidance

Exclusion Criteria:

• All other patients not list above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Video Consultations Completed | 1 year
  Total number of video consultations completed

SECONDARY OUTCOMES:
Mortality | 1 year
  Total number of subject deaths
Hospital Length of Stay | 1 year
  Total number of hours subjects were admitted to the hospital
Emergency Room Length of Stay | 1 year
  Total number of hours subjects were admitted to the emergency room

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Russi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials